CLINICAL TRIAL: NCT01736748
Title: Implementing Dynamo: a Tailored Lifestyle Promotion Intervention Among Pediatric Patients With Cardiometabolic Risk Factors
Brief Title: Dynamo: a Tailored Lifestyle Promotion Intervention Among Pediatric Patients With Cardiometabolic Risk Factors
Acronym: CIRCUIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Melanie Henderson, Endocrinologist and Assistant Clinical Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIRCUIT 1
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obese
Keywords: obesity; physical activity; metabolism; environment; obese children, as defined by a body mass index > 95th percentile; for age and sex
MeSH Terms: conditions — Obesity; Motor Activity; Coitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor based PA intervention (Experimental): Children will be equipped with a heart rate monitor, a GPS receiver and an accelerometer for collection of heart rate, mobility and physical activity free-living data during a 7-day period. This will provide a 'spatio-behavioural diagnosis' using a map-based interactive web application. This data will be used to developed a tailored plan to promote physical activity in the child's every day environment.
  Interventions: Behavioral: Sensor based PA intervention
- Traditional PA counseling (Other): In this arm, while children will wear the same sensors as in the intervention arm, the intervention will not rely on data gathered using the wearable sensors. Rather, a traditional physical activity counseling strategy will be adopted in this control group.
  Interventions: Behavioral: Traditional PA counseling

INTERVENTIONS:
Behavioral: Sensor based PA intervention — Children will be equipped with a heart rate monitor, a GPS receiver and an accelerometer for collection of heart rate, mobility and physical activity free-living data during a 7-day period. This will provide a 'spatio-behavioural diagnosis' using a map-based interactive web application. This data will be used to developed a tailored plan to promote physical activity in the child's every day environment.
  Arms: Sensor based PA intervention
Behavioral: Traditional PA counseling — Children will be encouraged to enhance their physical activity levels using traditional behavioral approaches.
  Arms: Traditional PA counseling

SUMMARY:
The Dyn@mo lifestyle intervention (CHU Sainte-Justine, Quebec, Canada) targets children and adolescents aged 6 to 17 years old with cardiometabolic risk factors, such as obesity, hypertension, disorders in glucose regulation or dyslipidemia. Its primary goal is to promote physical activity and reduce sedentary time to improve childrens' cardiometabolic profile. To do so, the intervention relies on gathering data on mobility and physical activity using wearable sensors. These data provide a detailed picture of real-life conditions and physical activity levels, improving the health care professional's ability to tailor counseling. The investigators are presently in the implementation phase of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* children ages 6 to 18 years of age with a BMI > 95th percentile for age and sex

Exclusion Criteria:

* children with a physical or psychological condition that would impair their ability to participate in physical activity

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity levels | Baseline and 1 year
  Physical activity will be measured using accelerometry and we will use time spent in moderate to vigorous physical activity as our primary measure of PA

SECONDARY OUTCOMES:
Change in blood pressure | Baseline and 1 year
  Both systolic and diastolic blood pressure will be measured
Change in glucose homeostasis | Baseline and 1 year
  Both fasting blood glucose, and glucose 2hr post load (oral glucose tolerance test) will be measured
Change in lipid status | Baseline and 1 year
  LDL, HDL, triglycerides and total cholesterol will be measured at baseline and after 1 year of follow-up
Change in body mass index | Baseline and 1 year
  We will measure height and weight at baseline and at 1 year of follow-up and calculate differences in body mass index over the 1 year period

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada